CLINICAL TRIAL: NCT04572126
Title: Feasibility and Efficacy of a Brief Mindfulness-Based Smoking Intervention Via the Internet
Brief Title: Feasibility and Efficacy of a Brief Mindfulness-Based Intervention SMOKING INTERVENTION VIA THE INTERNET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Michael Schmidt, Principal Investigator, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-20-09-2668
Record Dates: First submitted 2020-09-21; First posted 2020-10-01 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Substance Use; Smoking Reduction
Keywords: Smoking Reduction
MeSH Terms: conditions — Substance-Related Disorders; Smoking Reduction

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the mindfulness intervention group or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Group (Experimental): Participants in the mindfulness group will receive mindfulness based instructions.
  Interventions: Behavioral: Mindfulness Intervention
- Control Group (Active Comparator): Participants in the control group will receive instructions to cope with cravings how they normally would.
  Interventions: Behavioral: Control Intervention

INTERVENTIONS:
Behavioral: Mindfulness Intervention — The mindfulness intervention includes strategies to cope with substance cravings based on previously published mindfulness techniques. Examples of strategies presented include paying close attention to sensations, acceptance of cravings, and self-kindness.
  Arms: Mindfulness Group
Behavioral: Control Intervention — The control intervention instructs participants to utilize their own, previously used strategies to cope with substance cravings.
  Arms: Control Group

SUMMARY:
The current study will examine both the feasibility and efficacy of a single session, web-based mindfulness-based intervention for smoking cessation. The study will explore (1) participants' subjective experiences of the intervention, (2) cravings and negative affect both before and after the intervention, and (3) changes in tobacco use one week and one month following the initial intervention. Further, the study will examine how often participants utilize the intervention between the initial study and follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

* Daily Smoker
* Has a desire to quit or reduce smoking.
* Is not currently involved in another smoking reduction or cessation program.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Subjective Ratings Questionnaire | Immediately post-intervention
  The participant's ratings of subjective likeability and helpfulness of the intervention. These ratings will be measured on a 5-point Likert Scale with higher scores representing more likeability and helpfulness. The 11-item questionnaire results in a score ranging from 11-55.
Change in Past Month Cigarette and E-Cigarette use. | Immediately before the intervention and at one-month follow-up.
  An online version of the TLFB (Sobbel & Sobbel, 1992) will be used to measure past-month cigarette and e-cigarette use. The measure will be administered pre-intervention and one-month following the intervention to show change over time.
Change in Cigarette/E-cigarette Craving | Immediately preceding and following intervention.
  Craving to smoke will be measured using the 10-item Brief Questionnaire of Smoking Urges (Cox, Tiffany, & Christen, 2001).While the QSU-brief can be scored by using all 10 items for one total craving score, maximum likelihood factor analysis of the QSU-brief revealed a two-factor model consisting of (1) a strong desire and intention to smoke with the perception of receiving positive rewards from smoking and (2) the expectation that smoking would relieve negative affect and the strong desire to smoke. The measure will be administered immediately preceding and following the intervention to show intervention influence on craving.
Change in Positive and Negative Affect | Immediately preceding and following intervention as well as at one-month follow-up.
  Positive and negative affect will be measured by the Positive and Negative Affect Schedule (Watson & Clark, 1999).

SECONDARY OUTCOMES:
Intervention Use. | One-month after intervention.
  Number of times participants viewed intervention between intervention completion and one-month follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowen S, Marlatt A. Surfing the urge: brief mindfulness-based intervention for college student smokers. Psychol Addict Behav. 2009 Dec;23(4):666-71. doi: 10.1037/a0017127. PMID 20025372
- [Background] Brewer JA, Mallik S, Babuscio TA, Nich C, Johnson HE, Deleone CM, Minnix-Cotton CA, Byrne SA, Kober H, Weinstein AJ, Carroll KM, Rounsaville BJ. Mindfulness training for smoking cessation: results from a randomized controlled trial. Drug Alcohol Depend. 2011 Dec 1;119(1-2):72-80. doi: 10.1016/j.drugalcdep.2011.05.027. Epub 2011 Jul 1. PMID 21723049
- [Background] Witkiewitz K, Bowen S. Depression, craving, and substance use following a randomized trial of mindfulness-based relapse prevention. J Consult Clin Psychol. 2010 Jun;78(3):362-374. doi: 10.1037/a0019172. PMID 20515211